CLINICAL TRIAL: NCT00767988
Title: Probiotics Improvement of Gastrointestinal and Genitourinary Health in Girls With Spina Bifida (H-23245)
Brief Title: Probiotics in Girls With Spina Bifida
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn by PI
Sponsor: Baylor College of Medicine (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Eric A. Jones, M.D., Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-23245
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Urinary Tract Infection
Keywords: Probiotics; Spina Bifida; Dietary Supplements; Bacteriuria; Urinary Tract Infection (UTI)
MeSH Terms: conditions — Urinary Tract Infections; Spinal Dysraphism; Bacteriuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Urex-cap-5 capsules (2x10^9 cfu each of RC-14 and GR-1) 1:1 ratio
  Interventions: Dietary Supplement: Urex-cap-5 (2x10^9 cfu each of Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1)
- B (Placebo Comparator): Capsule 1:1
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Urex-cap-5 (2x10^9 cfu each of Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1) — Capsules once daily at approximately the same time each day for 6 months.
  Arms: A
Other: Placebo — Capsule once daily at approximately the same time each day for 6 months.
  Arms: B

SUMMARY:
Girls with spina bifida also have bladder problems. This is because they need temporary placement of a tube into the bladder to remove urine. This thin flexible tube is called a catheter. It can increase the risk of having bacteria in the urine. This in turn can lead to urinary tract infection (UTI).

Some girls with spina bifida are given antibiotics. These are medicines used to treat infections caused by bacteria. The medicine is used to prevent UTI. However, long-term treatment with these medicines can have side effects. For example, the bacteria may become resistant to the antibiotics. Also, bacteria in the urine can persist. UTI can still occur in patients on antibiotics.

UTI in girls occurs because bacteria migrate from the rectum to the vagina area. This gives the bacteria access to the bladder. Also, in girls with spina bifida, the access to the bladder is easier because of the catheter.

Probiotics are friendly bacteria. They are available as dietary supplements and as food. They contain helpful bacteria. Yogurt is an example of a food that contains probiotics.

The purpose of this study is to find out, if probiotics taken for 6 months can prevent UTI in girls with spina bifida. We will also try to find out whether changes in urine bacteria are associated with the taking of the probiotics. A vaginal and rectal swab will also be done to find out if taking probiotics has any benefits on preventing bacteria.

DETAILED DESCRIPTION:
In children with spina bifida and neurogenic bladder dysfunction, the need for intermittent bladder catheterization increases the risk of bacteriuria. In many patients, this leads to a clinically significant urinary tract infection (UTI). Many of these children are placed on long term, low dose antibiotic suppression to prevent recurrent urinary infection. Unfortunately, bacteriuria often persists despite daily antibiotic therapy, and breakthrough UTIs are common. Furthermore, this approach carries the potential for deleterious side effects, and may promote the development of antibiotic-resistant bacteria.

UTI in girls occur when virulent bacteria migrate from the rectum and colonize the vagina and peri-urethral mucosa, thus gaining access to the bladder. In girls with spina bifida, access to the bladder is greatly facilitated by catheter passage. Antibiotic prophylaxis relies on maintaining a low dose of antibiotic in the urinary stream, which decreases peri-urethral colonization, and prevents proliferation of bacteria after they gain access to the bladder. An alternative approach to daily antibiotic prophylaxis is to decrease the risk of urinary colonization with virulent bacteria by supplementing the normal bacteria flora with non-infection causing strains of bacteria.

Probiotics are dietary supplements containing potentially beneficial bacterial strains such as Lactobacillus. The safety of oral administration of probiotics has been demonstrated in several studies over the last 30 years. Studies using Lactobacillus rhamnosus GG, a probiotic introduced in the late 1980s to alleviate diarrhea, have shown promising results when used for UTI prevention. In one study, researchers found that the subjects consuming GG drinks had fewer episodes of UTI compared to those women not receiving probiotics. A placebo-controlled study in premature infants also used GG in an attempt to prevent UTI. The number of urinary infections was reduced but statistically the difference was not significant. Finally, a recent randomized clinical trial demonstrated that the rate of UTI in children taking prophylactic antibiotics was similar to that of patients taking Lactobacillus acidophilus alone. The efficacy of probiotic usage in the spina bifida population has not been reported.

Clinical trials have suggested that oral ingestion of the probiotic strains Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1 results in vaginal colonization and prevention of adult UTI, potentially by inhibiting uropathogen ascension from the vagina to the urinary tract.

A total of 60 patients will be enrolled for this pilot study, half of whom will be randomized to receive probiotics and the reminder of which will receive placebo [1:1 ratio; 50% chance of being in each group (A and B)]. Treatment assignment will be double blinded and will last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Girls
* Age 3 months to 18 years
* Spina bifida as a sole urologic diagnosis
* Informed consent and assent (7 years of age and older)

Exclusion Criteria:

* Males
* Females over 18 years and older
* Prophylactic antibiotics
* Immunosuppression from corticosteroids, transplant recipients or children with congenital immunodeficiencies
* Poorly controlled diabetes
* Untreated HIV infection
* Chronic indwelling catheters in the bladder
* Malnourished
* Pregnancy
* Any form of urinary division other than appendicovesicostomies is not permitted
* Bladder augmentation
* Unresolved reflux

Ages: 3 Months to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the rates of bacteriuria among patients in the placebo versus probiotics arms. | This will be calculated at the end of the 6 months of administering probiotics/placebo.

SECONDARY OUTCOMES:
The secondary outcomes include rates of fungal vaginitis, mean number of urinary tract infections, mean Bristol STool Scale scores, and number of episodes of stool incontinence. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric A. Jones, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - Shriner's Childrens Hospital Houston, Houston, Texas